CLINICAL TRIAL: NCT00127348
Title: Effect of CPAP on Arterial Hypertension and Cardiovascular Morbi-Mortality in Patients With Sleep Apnea and Without Daytime Sleepiness
Brief Title: Effect of Continuous Positive Airway Pressure (CPAP) on Hypertension and Cardiovascular Morbidity-Mortality in Patients With Sleep Apnea and no Daytime Sleepiness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI 040165
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2006-04

CONDITIONS: Sleep Apnea; Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypertension; Cardiovascular Diseases | interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Device: CPAP (Continuous Positive Airway Pressure)

SUMMARY:
The objective of the study is to evaluate the effect of CPAP over the incidence of cardiovascular events and diagnosis of arterial hypertension in patients with sleep apnea.

The hypothesis of the study is the following: The existence of sleep disordered breathing in the general population is associated to an increased incidence of arterial hypertension and to an increased risk of suffering cardiovascular disease. CPAP corrects respiratory disorders during sleep. Treatment with CPAP in subjects with sleep disordered breathing without daytime sleepiness reduces the incidence of systemic arterial hypertension and cardiovascular complications.

The end points of the study are new diagnosis of arterial hypertension and new cardiovascular events.

All patients, after randomization, will be followed for three years.

ELIGIBILITY:
Inclusion Criteria:

* Epworth <10
* Apnea-Hypopnea Index ≥20

Exclusion Criteria:

* Presence of any chronic disease
* Presence of cardiovascular disease
* Refusal to sign informed consent
* Drug addiction and/or alcoholism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 2004-05; Study Completion 2006-04

PRIMARY OUTCOMES:
Incidence of hypertension
Incidence of cardiovascular events

SECONDARY OUTCOMES:
Relationship between hypertension and sleep apnea/hypopnea syndrome (SAHS) severity
Relationship between cardiovascular events and SAHS severity

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbe, MD, Principal Investigator — Hospital Universitari Arnau de Vilanova. Lleida. Spain
Locations (1):
- Hospital Univ Arnau de Vilanova, Lleida, Catalonia, Spain

REFERENCES:
- [Derived] Reynor A, McArdle N, Shenoy B, Dhaliwal SS, Rea SC, Walsh J, Eastwood PR, Maddison K, Hillman DR, Ling I, Keenan BT, Maislin G, Magalang U, Pack AI, Mazzotti DR, Lee CH, Singh B. Continuous positive airway pressure and adverse cardiovascular events in obstructive sleep apnea: are participants of randomized trials representative of sleep clinic patients? Sleep. 2022 Apr 11;45(4):zsab264. doi: 10.1093/sleep/zsab264. PMID 34739082
- [Derived] Phillips B, Shafazand S. CPAP and hypertension in nonsleepy patients. J Clin Sleep Med. 2013 Feb 1;9(2):181-2. doi: 10.5664/jcsm.2426. PMID 23372475
- [Derived] Weaver TE, Mancini C, Maislin G, Cater J, Staley B, Landis JR, Ferguson KA, George CF, Schulman DA, Greenberg H, Rapoport DM, Walsleben JA, Lee-Chiong T, Gurubhagavatula I, Kuna ST. Continuous positive airway pressure treatment of sleepy patients with milder obstructive sleep apnea: results of the CPAP Apnea Trial North American Program (CATNAP) randomized clinical trial. Am J Respir Crit Care Med. 2012 Oct 1;186(7):677-83. doi: 10.1164/rccm.201202-0200OC. Epub 2012 Jul 26. PMID 22837377
- [Derived] Barbe F, Duran-Cantolla J, Sanchez-de-la-Torre M, Martinez-Alonso M, Carmona C, Barcelo A, Chiner E, Masa JF, Gonzalez M, Marin JM, Garcia-Rio F, Diaz de Atauri J, Teran J, Mayos M, de la Pena M, Monasterio C, del Campo F, Montserrat JM; Spanish Sleep And Breathing Network. Effect of continuous positive airway pressure on the incidence of hypertension and cardiovascular events in nonsleepy patients with obstructive sleep apnea: a randomized controlled trial. JAMA. 2012 May 23;307(20):2161-8. doi: 10.1001/jama.2012.4366. PMID 22618923
- [Derived] Barbe F, Duran-Cantolla J, Capote F, de la Pena M, Chiner E, Masa JF, Gonzalez M, Marin JM, Garcia-Rio F, de Atauri JD, Teran J, Mayos M, Monasterio C, del Campo F, Gomez S, de la Torre MS, Martinez M, Montserrat JM; Spanish Sleep and Breathing Group. Long-term effect of continuous positive airway pressure in hypertensive patients with sleep apnea. Am J Respir Crit Care Med. 2010 Apr 1;181(7):718-26. doi: 10.1164/rccm.200901-0050OC. Epub 2009 Dec 10. PMID 20007932